CLINICAL TRIAL: NCT06411197
Title: Exploration of Gait Biomechanics and Muscle Pain of the Lower Extremity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kristian Kjær Petersen (Other)
Responsible Party: Sponsor-Investigator, Kristian Kjær Petersen, Associate professor, Aalborg University
Organization: Aalborg University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20220063-2
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Pain, Acute
Keywords: Musculoskeletal pain; Healthy Participants; Biomechanics
MeSH Terms: conditions — Acute Pain; Musculoskeletal Pain | interventions — Saline Solution, Hypertonic; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Gastrocnemius (painful condition) (Experimental): 1.5 mL injection of hypertonic saline (7%) to the gastrocnemius muscle.
  Interventions: Other: Hypertonic saline injection
- Gastrocnemius (control condition) (Sham Comparator): 1.5 mL injection of isotonic saline (0.9%) to the gastrocnemius muscle.
  Interventions: Other: Isotonic saline injection
- Biceps femoris (painful condition) (Experimental): 1.2 mL injection of hypertonic saline (7%) to the biceps femoris muscle.
  Interventions: Other: Hypertonic saline injection
- Biceps femoris (control condition) (Sham Comparator): 1.2 mL injection of isotonic saline (0.9%) to the biceps femoris muscle.
  Interventions: Other: Isotonic saline injection
- Semitendinosus (painful condition) (Experimental): 1.2 mL injection of hypertonic saline (7%) to the semitendinosus muscle.
  Interventions: Other: Hypertonic saline injection
- Semitendinosus (control condition) (Sham Comparator): 1.2 mL injection of isotonic saline (7%) to the semitendinosus muscle.
  Interventions: Other: Isotonic saline injection

INTERVENTIONS:
Other: Hypertonic saline injection — Injection with hypertonic saline (7%)
  Arms: Biceps femoris (painful condition); Gastrocnemius (painful condition); Semitendinosus (painful condition)
Other: Isotonic saline injection — Injection with isotonic saline (0.9%)
  Arms: Biceps femoris (control condition); Gastrocnemius (control condition); Semitendinosus (control condition)

SUMMARY:
This interventional study aims to test gait biomechanics in healthy individuals with and without experimental muscle pain in the lower extremities. The study aims to:

A) Examine how experimental muscle pain in different types of muscles (ankle plantar-flexion, knee extension, and flexion muscles) affects kinematics, kinetics, and muscle activation

Participants will receive six muscle injections: a) Hypertonic saline (painful condition) and b) Isotonic saline (control condition) in 1) m. gastrocnemius, 2) m. semitendinosus, and 3) m. biceps femoris.

DETAILED DESCRIPTION:
The proposed study will be a randomized, crossover design in which experimental pain will be induced in healthy subjects using hypertonic saline injections to three muscles of the lower extremities: The gastrocnemius muscle, the vastus medialis muscle, and the semitendinosus muscle. Participants will be block-randomized to receive an injection in each of the three muscles and will receive either the painful or control condition first for each muscle. The participant will always be blinded to the type of injection received.

Following the injection, there will typically be a 15-minute window of pain (45). Within this timeframe, motion capture will be carried out for both the control and painful conditions. During motion capture, the participants will perform multiple walking trials of approximately 10 meters. The participants will be equipped with electromyography (EMG) sensors on key muscles of the lower extremities. The participants will be asked for NRS ratings every 30 seconds throughout the 15 minutes with expected pain. There will be a 15-minute washout between the muscle injections.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 18-45 years

Exclusion Criteria:

* Pregnancy
* Drug addiction, defined as the use of cannabis, opioids, or other drugs
* Previous or current neurologic or musculoskeletal illnesses
* Current pain
* Lack of ability to cooperate

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Infrared marker XYZ coordinates | Baseline.
  Marker-based motion capture with infrared cameras will be used to estimate placement of reflective markers in the XYZ planes measured in millimeters. Reflective markers will be placed from head-to-toe on anatomical landmarks.
Pain intensity (NRS 0-10) | Baseline.
  Pain during intervention is measured continuously every 30 seconds on a numeric rating scale from 0 'no pain' to 10 'the worst pain imaginable'

SECONDARY OUTCOMES:
Pain sensitivity. | Baseline.
  Cuff-pressure algometry will be used to estimate pressure detection and tolerance thresholds, temporal summation of pain, and conditioned pain modulation.
Ground reaction forces | Baseline.
  Ground reaction forces will be measured in Newtons with force plates embedded in the floor.
Ground reaction moments | Baseline.
  Ground reaction moments will be measured in Newton-meters with force plates embedded in the floor.
Ground contact XZ location | Baseline.
  Ground contact XZ coordinate location will be measured in millimeters with force plates embedded in the floor.
Muscle activation | Baseline.
  Muscle activation will be measured in micro-volts using wireless EMG on the muscles of the lower extremities.

OTHER OUTCOMES:
Pain during jumping | Baseline
  Pain during jumping is captured on a numeric rating scale from 0 'no pain' to 10 'the worst pain imaginable'

CONTACTS AND LOCATIONS:
Overall Officials: Kristian KS Petersen, Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided